CLINICAL TRIAL: NCT00942318
Title: Efficacy of Continuous Subcutaneous Insulin Infusion Versus Basal-bolus Multiple Daily Injections Regimen in Type 2 Diabetes: a One Year, Randomised, Parallel Study
Brief Title: Efficacy of Continuous Subcutaneous Insulin Infusion Versus Basal-bolus Multiple Daily Injections Regimen in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0816202; AOL 2008
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Continuous subcutaneous insulin infusion; Insulin external pump; Multiple daily injections; Basal-bolus regimen; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPE (Experimental): PPE : CSII +/- Metformin.
  Interventions: Drug: Detemir insulin, Aspart insulin, Metformin
- injections (Active Comparator): INJ: basal/bolus MDI +/- Metformin
  Interventions: Drug: Detemir insulin, Aspart insulin, Metformin

INTERVENTIONS:
Drug: Detemir insulin, Aspart insulin, Metformin — Insulin doses adapted by patients according to self monitoring blood glucose results.

SUMMARY:
A lot of insulin-treated type 2 diabetic patients do not reach adequate glycemic control despite intensive basal-bolus insulin regimen. In such cases, continuous subcutaneous insulin infusion (CSII), using an external pump, could be a solution to improve diabetes control.

The aim of this study is to compare, over a one-year period, the efficacy of CSII (with aspart insulin) and basal-bolus multiple daily injections (MDI) treatment (with detemir x 2/d and aspart before meals) in type 2 diabetic patients, already treated by basal-bolus regimen for at least 6 months, who didn't reach adequate target for glycemic at baseline (HbA1c>7 -10%).

DETAILED DESCRIPTION:
Visit 1: patient information and eligibility criteria assessment Visit 2: Inform consent signature and randomisation (group CSII or MDI). Patients randomised in the CSII group are instructed to use pump between V2 and V3.

Visit 3: 5-day's hospitalisation. Start of CSII or MDI treatments. Stop of all oral diabetic medications except for metformin, which is followed up until the end of the study. Teaching program on diabetes management (diet, physical activity and self-adjustment of insulin doses). HbA1c, clinical and biological parameters. Questionnaires.

Follow-up visits 4-7 (1, 3, 6, 9 months): HbA1c. Treatment adjustment. Adverse events collection.

Final visit (12 months): HbA1c, clinical and biological parameters. Questionnaires. Adverse events collection.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Age > 18 years
* Patients treated for at least 6 months by Multiple daily insulin injections associating long acting insulin (at least 1 long acting insulin analog injection -Glargine or Detemir- or at least 2 NPH insulin injections) plus mealtimes rapid acting insulin injections (Human or analogs) +/- oral hypoglycemic agents.
* 7,5% ≤ HbA1c ≤ 10%
* Patients able to perform self-monitoring blood glucose (SMBG) measurement and insulin injections.
* SMBG > 3/day

Exclusion Criteria:

* Diabetic retinopathy contraindicating glycemic control intensification
* Situation or pathology not allowing therapeutic education program (blindness, deafness, low language fluency…)
* Situation or pathology not allowing insulin therapy self-management and / or portable insulin pump use (rheumatologic pathology, low visual acuity, …)
* Recent (<3 month) serious pathology
* Planned treatment or therapy able to induce long-term glycemic control worsening
* Long lasting (> 2 month) planned treatment with glucocorticoids, octreotide, lanreotide or danazol
* Pregnancy wish or ongoing pregnancy
* Known Haemoglobinopathy.
* Creatinin clearance <30ml/min (MDRD formula).
* Organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months

SECONDARY OUTCOMES:
Weight, waist perimeter, BP, triglycerides, total cholesterol, HDL and LDL cholesterol ; QOL, physical activity, treatment satisfaction and eating habits questionnaire. | 12 months
self monitoring blood glucose measurements (frequency, mean and standard deviation, number of hypoglycaemic and hyperglycaemic events) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Melki, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France